CLINICAL TRIAL: NCT00336882
Title: Anaesthesia With Propofol Versus Midazolam : Effect on Oxidative Stress in the Brain of Head Trauma Patients
Acronym: PROMIS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EUDRACT 2005-006213-40; PHRC/05-02 (Other: Rennes University Hospital); CIC0203/053
Record Dates: First submitted 2006-06-13; First posted 2006-06-14 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; propofol; oxidative stress; microdialysis
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Propofol; Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Midazolam at a dose of 0,03 mg/kg/hour with dose increasing of 0,02 mg/kg/hour until therapeutic effect.
  Interventions: Drug: Midazolam
- 2 (Experimental): Propofol at a dose of 1 mg/kg/hour with a dose increase of 1 mg/kg until therapeutic effect (with a maximum dose of 5 mg/kg/hour)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol at a dose of 1 mg/kg/hour with a dose increase of 1 mg/kg until therapeutic effect (with a maximum dose of 5 mg/kg/hour)
  Other Names: DIPRIVAN
  Arms: 2
Drug: Midazolam — Midazolam at a dose of 0,03 mg/kg/hour with dose increasing of 0,02 mg/kg/hour until therapeutic effect.
  Other Names: HYPNOVEL
  Arms: 1

SUMMARY:
Severe traumatic brain injury is associated with an increased production of free radicals causing brain damage. First line treatment of these patients aims to maintain cerebral perfusion and includes deep anaesthesia. Propofol has recently shown anti oxidant properties that need to be confirmed when used in these patients. The main objective of this study is to evaluate the effect of propofol compared to midazolam on intra cerebral oxidative stress following severe traumatic brain injury.

DETAILED DESCRIPTION:
Severe traumatic brain injury is associated with an increased production of free radicals causing brain damage. First line treatment of these patients aims to maintain cerebral perfusion and includes deep anaesthesia. Propofol has recently shown anti oxidant properties that need to be confirmed when used in these patients. The main objective of this study is to evaluate the effect of propofol compared to midazolam on intra cerebral oxidative stress following severe traumatic brain injury. Measurements will be performed by use of intracerebral microdialysis.

ELIGIBILITY:
Inclusion Criteria:

Age≥18 years, Severe traumatic brain injury with a Glasgow coma scale ≤8 related to the trauma, Stage II, III or IV of the US Trauma Data Bank on the CT scan, Need for intracranial pressure monitoring, Written informed consent from the patient's next-of-kin. If no relative is present as the time of inclusion, the patients will be included according to the emergency procedure.

Non-inclusion Criteria:

Traumatic brain injury requiring urgent neurosurgical intervention due to blood collection, Contraindication to propofol or midazolam, History of head trauma > 12 hours before intra cranial pressure monitoring, Patient receiving propofol by continuous infusion since head trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-06; Primary Completion 2009-10 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Lactate/pyruvate ratio concentration measured in the brain by microdialysis during the first 72 h of treatment | 72 hours

SECONDARY OUTCOMES:
Glutamate, glucose and glycerol concentration measured in the brain by microdialysis during the first 72 h of treatment. | 72 hours
Glasgow outcome scale and Mc Nair score at 12 months. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Mallédant, MD, PhD, Principal Investigator — Rennes University Hospital; Bruno Laviolle, MD, Study Chair — Rennes University Hospital
Locations (1):
- Réanimation Chirurgicale - Hôpital de Pontchaillou, Rennes, France